CLINICAL TRIAL: NCT02400476
Title: An Open-Label Study to Characterize the Incidence and Severity of Diarrhea in Patients With Early-Stage HER2+ Breast Cancer Treated With Neratinib and Loperamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PUMA-NER-6201; 2015-004374-15 (EudraCT Number)
Record Dates: First submitted 2015-02-17; First posted 2015-03-27 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-01

CONDITIONS: Early Stage HER2+ Breast Cancer
Keywords: HER2 +; Breast Cancer; Neratinib; Nerlynx; Loperamide; Colestipol; Budesonide
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Loperamide; Colestipol; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Loperamide (Experimental): 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Loperamide daily for two 28-day cycles and then as needed.
  Interventions: Drug: Neratinib; Drug: Loperamide
- Budesonide and Loperamide (Experimental): 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Anti-inflammatory treatment for 1 cycle and Loperamide to be administered daily for two 28-day cycles and then as needed, thereafter.
  Interventions: Drug: Neratinib; Drug: Loperamide; Drug: Budesonide
- Colestipol and Loperamide (Experimental): 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Colestipol for 1 cycle and loperamide to be administered 1 cycle and then as needed, thereafter.
  Interventions: Drug: Neratinib; Drug: Loperamide; Drug: Colestipol
- Colestipol with Loperamide as needed (Experimental): 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Colestipol for 1 cycle and loperamide to be administered as needed.
  Interventions: Drug: Neratinib; Drug: Loperamide; Drug: Colestipol
- Neratinib Dose Escalation 1 (Experimental): 120 mg Neratinib for Week 1, followed by 160 mg Neratinib starting for Week 2, followed by 240 mg Neratinib starting at Week 3 and thereafter (C1D15 to End of Treatment). Loperamide administered as needed.
  Interventions: Drug: Neratinib; Drug: Loperamide
- Neratinib Dose Escalation 2 (Experimental): 160 mg neratinib for the first 2 weeks, followed by 200 mg neratinib for the next 2 weeks, followed by 240 mg neratinib thereafter (C2D1 to End of treatment. Loperamide will be administered on an as-needed basis only.
  Interventions: Drug: Neratinib; Drug: Loperamide

INTERVENTIONS:
Drug: Neratinib
  Other Names: Nerlynx
Drug: Loperamide
Drug: Colestipol — 2 g twice daily with or without food for one 28 day cycle
  Arms: Colestipol and Loperamide; Colestipol with Loperamide as needed
Drug: Budesonide — 9 mg extended release tablets once daily with or without food for 28 days
  Arms: Budesonide and Loperamide

SUMMARY:
An Open-Label Study to Characterize the Incidence and Severity of Diarrhea in Patients with Early-Stage HER2+ Breast Cancer Treated with Neratinib and Loperamide or other prophylactic measures.

DETAILED DESCRIPTION:
This is an open-label, Phase 2 study that will investigate the incidence and severity of diarrhea in early-stage HER2+ breast cancer patients receiving neratinib with loperamide, alone and in combination with an anti-inflammatory treatment or a bile acid sequestrant treatment, or neratinib dose escalation, who have previously undergone a course of trastuzumab therapy in the adjuvant setting.

Patients will receive:

* Neratinib 240 mg orally once daily with food for thirteen 28-day cycles.
* Loperamide daily for two 28-day cycles and then as needed.
* Amendment 3, an anti-inflammatory treatment for one cycle and loperamide to be administered daily for two 28-day cycles and then as needed. Closed to enrollment.
* Amendment 4, colestipol for one cycle and loperamide to be administered one cycle and then as needed. Closed to enrollment.
* Amendment 5, colestipol for one cycle and loperamide as needed. Closed to enrollment.
* Amendment 6/6.1, 120 mg neratinib for Week 1 (C1D1-C1D7), followed by 160 mg neratinib for Week 2 (C1D8-C1D14), followed by 240 mg neratinib for Week 3 and thereafter (C1D15 to end of treatment). Loperamide as needed. Closed to enrollment.
* Amendment 7/7.1, 160 mg neratinib for the first 2 weeks (C1D1 - C1D14), followed by 200 mg neratinib for the next 2 weeks (C1D15 - C1D28), followed by 240 mg neratinib thereafter (C2D1 to end of treatment). Loperamide as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18; male or female
* Early breast cancer (stage I-3c)
* Documented HER2+ tumor: HER2 immunohistochemistry (IHC) 3+ or ISH+
* Prior course of adjuvant trastuzumab given >2 weeks and ≤1 year from enrollment
* No evidence of local/regional recurrence or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Male patients with female partners of childbearing potential must agree and commit to use a condom and women of childbearing potential must not be pregnant and must agree and commit to the use of a highly effective non-hormonal method of contraception
* Left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or ECHO

Exclusion Criteria:

* Major surgery < 30 days
* Chemotherapy, investigational agents, other cancer therapy (except hormonal therapy) < 14 days
* Corrected QT Interval (QTc) >0.450 seconds (males) or >0.470 (females) or other active cardiac disease
* Significant chronic GI disorder with diarrhea as a major symptom
* Active, unresolved infections
* Currently pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Puma Biotechnology, Inc.
Locations (58):
- United States (39):
  - Alabama Oncology, Birmingham, Alabama
  - Compassionate Care Research Group Inc., Corona, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Emad Ibrahim, M.D., Inc., Redlands, California
  - Torrance Memorial Physician Network Cancer Care Associates, Redondo Beach, California
  - Compassionate Care Research Group Inc., Riverside, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - Cancer Center of Santa Barbara with Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Memorial Healthcare System, Hollywood, Florida
  - Florida Cancer Research Institute, LLC, Plantation, Florida
  - Hematology-Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Baptist Health Urgent Care Sawgrass, Sunrise, Florida
  - Cancer Treatment Centers of America, Newnan, Georgia
  - Decatur Memorial Hospital Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Central Maine Medical Center, Lewiston, Maine
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - North Mississippi Medical Center Hematology and Oncology Services, Tupelo, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Great Plains Health (Callahan Cancer Center), North Platte, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey
  - Clinical Research Alliance, Inc, Lake Success, New York
  - Good Samaritan Hospital Samaritan Pastega Regional Cancer Center, Corvallis, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Saint Joseph / Candler SC Cancer Specialists, Hilton Head Island, South Carolina
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Australia (3):
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - BCRC-WA, Hollywood Private Hospital, Nedlands, Western Australia
- Austria (5):
  - Univ. Klinik für Innere Medizin, Klin. Abt. Onkologie, Graz
  - Medical University of Innsbruck-Department of Gynecology, Innsbruck
  - Uniklinikum Salzburg, Landeskrankenhaus, Univ. Klinik fur Innere Medizin III der PMU, Salzburg
  - Medical University of Vienna, Department of Oncology, Vienna
  - Medical University of Vienna,Department of Obstetrics and Gynecology, Vienna
- Canada (2):
  - Sunnybrook Research Insitute, Toronto, Ontario
  - McGill University Health Centre, Cedars Cancer Centre, Montreal, Quebec
- France (2):
  - CHU Group Hospitalier Pitié-Salpêtrière, Service d'oncologie Médicale, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Schleswig-Holstein (UKSH), Klinik fuer Gynaekologie und Geburtshilfe, Studienzentrale Gynäkologische Onkologie (SGC) Kiel, Kiel
  - Sana Klinikum Offenbach GmbH - Frauenklinik, Offenbach
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://www.pumabiotechnology.com/data_sharing_policy.html

REFERENCES:
- [Derived] Chan A, Ruiz-Borrego M, Marx G, Chien AJ, Rugo HS, Brufsky A, Thirlwell M, Trudeau M, Bose R, Garcia-Saenz JA, Egle D, Pistilli B, Wassermann J, Cheong KA, Schnappauf B, Semsek D, Singer CF, Foruzan N, DiPrimeo D, McCulloch L, Hurvitz SA, Barcenas CH. Final findings from the CONTROL trial: Strategies to reduce the incidence and severity of neratinib-associated diarrhea in patients with HER2-positive early-stage breast cancer. Breast. 2023 Feb;67:94-101. doi: 10.1016/j.breast.2022.12.003. Epub 2022 Dec 14. PMID 36702070
- [Derived] Barcenas CH, Hurvitz SA, Di Palma JA, Bose R, Chien AJ, Iannotti N, Marx G, Brufsky A, Litvak A, Ibrahim E, Alvarez RH, Ruiz-Borrego M, Chan N, Manalo Y, Kellum A, Trudeau M, Thirlwell M, Garcia Saenz J, Hunt D, Bryce R, McCulloch L, Rugo HS, Tripathy D, Chan A; CONTROL Study Investigators. Improved tolerability of neratinib in patients with HER2-positive early-stage breast cancer: the CONTROL trial. Ann Oncol. 2020 Sep;31(9):1223-1230. doi: 10.1016/j.annonc.2020.05.012. Epub 2020 May 25. PMID 32464281

RESULTS

PARTICIPANT FLOW:
Groups:
- Loperamide: 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Loperamide daily for two 28-day cycles and then as needed.
  Neratinib
  Loperamide
- Budesonide and Loperamide: 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Anti-inflammatory treatment for 1 cycle and Loperamide to be administered daily for two 28-day cycles and then as needed, thereafter.
  Neratinib
  Loperamide
  Budesonide: 9 mg extended release tablets once daily with or without food for 28 days
- Colestipol and Loperamide: 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Colestipol for 1 cycle and loperamide to be administered 1 cycle and then as needed, thereafter.
  Neratinib
  Loperamide
  Colestipol: 2 g twice daily with or without food for one 28 day cycle
- Colestipol With Loperamide as Needed: 240 mg Neratinib orally once daily with food for thirteen 28-day cycles. Colestipol for 1 cycle and loperamide to be administered as needed.
  Neratinib
  Loperamide
  Colestipol: 2 g twice daily with or without food for one 28 day cycle
- Neratinib Dose Escalation 1: 120 mg Neratinib for Week 1, followed by 160 mg Neratinib starting for Week 2, followed by 240 mg Neratinib starting at Week 3 and thereafter (C1D15 to End of Treatment). Loperamide administered as needed.
  Neratinib
  Loperamide
- Neratinib Dose Escalation 2: 160 mg neratinib for the first 2 weeks, followed by 200 mg neratinib for the next 2 weeks, followed by 240 mg neratinib thereafter (C2D1 to End of treatment. Loperamide will be administered on an as-needed basis only.
  Neratinib
  Loperamide
Period: Overall Study
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2
Started | 137 | 64 | 136 | 104 | 60 | 62
Completed | 76 | 52 | 95 | 74 | 45 | 46
Not Completed | 61 | 12 | 41 | 30 | 15 | 16
Not completed — Adverse Event | 57 | 10 | 22 | 19 | 5 | 8
Not completed — Withdrawal by Subject | 4 | 1 | 12 | 7 | 5 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Other, Disease Progression | 0 | 1 | 2 | 1 | 2 | 1
Not completed — Other, Decreased Quality of Life | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other, Noncompliance to Protocol Requirements | 0 | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2 | Total
Number analyzed (Participants) | 137 | 64 | 136 | 104 | 60 | 62 | 563
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 116 | 58 | 117 | 93 | 51 | 52 | 487
  >=65 years | 21 | 6 | 19 | 11 | 9 | 10 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.39 (11.06) | 49.11 (10.55) | 52.49 (11.08) | 51.94 (10.23) | 51.90 (10.71) | 53.82 (10.15) | 52.31 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 64 | 133 | 104 | 60 | 62 | 560
  Male | 0 | 0 | 3 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 113 | 50 | 96 | 80 | 53 | 52 | 444
  Race: Black or African American | 11 | 5 | 9 | 8 | 1 | 2 | 36
  Race: Asian | 8 | 4 | 13 | 9 | 3 | 1 | 38
  Race: American Indian or Alaska Native | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 3 | 0 | 0 | 0 | 4
  Race: Other | 3 | 2 | 9 | 0 | 1 | 3 | 18
  Race: Unknown | 0 | 1 | 2 | 1 | 0 | 1 | 5
  Race: Missing | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Race: Not Reported | 1 | 1 | 3 | 6 | 2 | 2 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 4 | 10 | 6 | 7 | 27
  Austria | 0 | 0 | 0 | 0 | 0 | 4 | 4
  United States | 132 | 52 | 115 | 83 | 20 | 11 | 413
  Australia | 5 | 12 | 17 | 11 | 23 | 18 | 86
  France | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Germany | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Spain | 0 | 0 | 0 | 0 | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Grade 3 or Higher Diarrhea, According to NCI CTCAE v4.0.
Description: The primary objective of this study is to characterize the percentage of patients with Grade 3 or higher diarrhea in patients with early-stage HER2 overexpressed/amplified (HER2+) breast cancer treated with neratinib when administered with intensive loperamide prophylaxis, after prior treatment with trastuzumab. Grade 3: Increase of >=7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death.
Time Frame: From first dose of investigational product through 28 days after last dose, up to 15.5 months.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2
Number analyzed (Participants) | 137 | 64 | 136 | 104 | 60 | 62
Percentage of participants | 30.7 [23.1 to 39.1] | 28.1 [17.6 to 40.8] | 20.6 [14.1 to 28.4] | 32.7 [23.8 to 42.6] | 13.3 [5.9 to 24.6] | 27.4 [16.9 to 40.2]

2. Secondary Outcome: Percentage of Patients With Diarrhea by Grade, According to the National Cancer Institute Common Terminology Criteria (NCI CTCAE), Version 4.0.
Description: Assess the percentage of patients with diarrhea after the administration of an anti-inflammatory agent, a bile acid sequestrant, or following two different dose-escalation regimens of neratinib, by maximum CTC grade. Grade 1: an increase of <4 stools per day over baseline; mild increase in ostomy output compared to baseline. Grade 2: Increase of 4 - 6 stools per day over baseline; moderate increase in ostomy output compared to baseline. Grade 3: Increase of >=7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared to baseline; limiting self care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death.
Time Frame: From first dose of investigational product through 28 days after last dose, up to 15.5 months.
Measure: Number; unit: Percentage of participants
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2
Number analyzed (Participants) | 137 | 64 | 136 | 104 | 60 | 62
Percentage of participants
  Percentage of Patients w Grade 1 Diarrhea | 24.1 | 23.4 | 27.9 | 32.7 | 40.0 | 37.1
  Percentage of Patients w Grade 2 Diarrhea | 24.8 | 34.4 | 34.6 | 29.8 | 45.0 | 33.9
  Percentage of Patients w Grade 3 Diarrhea | 30.7 | 28.1 | 20.6 | 32.7 | 13.3 | 27.4

3. Secondary Outcome: Percentage of Patients With Serious Adverse Events and Other Adverse Events of Special Interest
Description: Assess the percentage of patients with serious adverse events (SAEs) and other adverse events of special interest (AESI). AESIs were selected based on the known safety profile of neratinib as well as typical key body system toxicity concerns generally reviewed for any new drug. These AESIs were grouped into the following categories: gastrointestinal toxicity (diarrhea and stomatitis), hepatotoxicity, pulmonary toxicity (interstitial lung disease), cardiac toxicity (LVEF decreased), and dermatologic toxicity (rash and nail disorders). The AESIs were analyzed by searching the clinical database for all TEAEs and SAEs using either Standardized MedDRA Queries (SMQs) or, if an applicable SMQ did not exist, a Sponsor-defined list of MedDRA preferred terms.
Time Frame: From first dose of investigational product through 28 days after last dose, up to 15.5 months.
Population: All subjects who received at least one dose of neratinib.
Measure: Number; unit: percentage of participants
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2
Number analyzed (Participants) | 137 | 64 | 136 | 104 | 60 | 62
percentage of participants
  Percentage of Patients with SAEs | 6.57 | 6.25 | 6.62 | 2.88 | 8.33 | 8.06
  Percentage of Patients with AESI-Gastrointestinal Toxicities (Diarrhoea and Stomatitis Broad Search) | 81.75 | 87.5 | 83.82 | 96.15 | 98.33 | 98.39
  Percentage of Patients with-Hepatotoxicities SMQ (Broad Search) | 12.41 | 7.81 | 4.41 | 4.81 | 8.33 | 4.84
  Percentage of Patients with AESI- Interstitial Lung Disease SMQ (Broad Search) | 0 | 0 | 0 | 0 | 0 | 0
  Percentage of Patients with AESI-Cardiac Toxicities SMQ (Broad Search) | 5.84 | 6.25 | 10.29 | 7.69 | 10.00 | 4.84
  Percentage of Patients with AESI - Dermatologic Toxicities (Rash and Nail Disorders) | 12.41 | 37.50 | 23.53 | 18.27 | 11.67 | 30.65
  Percentage of Patients with AESI-Gastrointestinal Toxicities (Narrow Search) | 80.29 | 85.94 | 83.09 | 95.19 | 98.33 | 98.39
  Percentage of Patients with AESI-Hepatotoxicities SMQ (Narrow Search) | 10.95 | 7.81 | 3.68 | 3.85 | 8.33 | 4.84
  Percentage of Patients with AESI- Interstitial Lung Disease SMQ (Narrow Search) | 0 | 0 | 0 | 0 | 0 | 0
  Percentage of Patients with AESI-Cardiac Toxicities SMQ (Narrow Search) | 2.92 | 0 | 1.47 | 0.96 | 1.67 | 0

ADVERSE EVENTS:
Time Frame: From time of first dose, through 28 days after last dose, assessed up to 15.5 months.
Arm/Group | Loperamide | Budesonide and Loperamide | Colestipol and Loperamide | Colestipol With Loperamide as Needed | Neratinib Dose Escalation 1 | Neratinib Dose Escalation 2
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/64 | 0/136 | 0/104 | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 9/137 | 4/64 | 9/136 | 3/104 | 5/60 | 5/62
Other Adverse Events (participants affected / at risk) | 137/137 | 64/64 | 136/136 | 104/104 | 60/60 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loperamide (N=137) | Budesonide and Loperamide (N=64) | Colestipol and Loperamide (N=136) | Colestipol With Loperamide as Needed (N=104) | Neratinib Dose Escalation 1 (N=60) | Neratinib Dose Escalation 2 (N=62)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fat necrosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Loperamide (N=137) | Budesonide and Loperamide (N=64) | Colestipol and Loperamide (N=136) | Colestipol With Loperamide as Needed (N=104) | Neratinib Dose Escalation 1 (N=60) | Neratinib Dose Escalation 2 (N=62)
Anaemia (Blood and lymphatic system disorders) | 8 | 5 | 1 | 5 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 4 | 3 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 7 | 2 | 7 | 5 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 21 | 5 | 22 | 15 | 6 | 10
Abdominal pain (Gastrointestinal disorders) | 36 | 12 | 26 | 27 | 13 | 15
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 16 | 7 | 3 | 8
Constipation (Gastrointestinal disorders) | 78 | 48 | 93 | 39 | 22 | 15
Diarrhoea (Gastrointestinal disorders) | 109 | 55 | 113 | 99 | 59 | 61
Dry mouth (Gastrointestinal disorders) | 18 | 6 | 12 | 5 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 12 | 10 | 16 | 13 | 7 | 6
Flatulence (Gastrointestinal disorders) | 5 | 6 | 5 | 2 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 5 | 10 | 6 | 2 | 4
Nausea (Gastrointestinal disorders) | 78 | 32 | 83 | 64 | 27 | 28
Stomatitis (Gastrointestinal disorders) | 7 | 4 | 14 | 13 | 6 | 6
Vomiting (Gastrointestinal disorders) | 36 | 16 | 43 | 25 | 9 | 5
Asthenia (General disorders) | 6 | 1 | 1 | 4 | 3 | 2
Fatigue (General disorders) | 73 | 34 | 65 | 41 | 28 | 19
Pyrexia (General disorders) | 6 | 2 | 10 | 3 | 2 | 1
Cellulitis (Infections and infestations) | 3 | 1 | 0 | 2 | 3 | 0
Influenza (Infections and infestations) | 2 | 0 | 3 | 4 | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 2 | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 7 | 7 | 5 | 6 | 2
Urinary tract infection (Infections and infestations) | 10 | 2 | 8 | 9 | 6 | 5
Alanine aminotransferase increased (Investigations) | 9 | 4 | 4 | 3 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 3 | 2 | 3 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 10 | 4 | 11 | 4 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 26 | 11 | 24 | 26 | 8 | 8
Dehydration (Metabolism and nutrition disorders) | 7 | 6 | 5 | 4 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 8 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 14 | 15 | 13 | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 5 | 9 | 10 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 8 | 14 | 15 | 12 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 6 | 5 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 7 | 5 | 2 | 3
Dizziness (Nervous system disorders) | 19 | 6 | 21 | 20 | 9 | 8
Headache (Nervous system disorders) | 26 | 12 | 20 | 24 | 13 | 8
Neuropathy peripheral (Nervous system disorders) | 4 | 3 | 3 | 6 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 1 | 3 | 0 | 5 | 0
Anxiety (Psychiatric disorders) | 5 | 4 | 3 | 3 | 3 | 2
Insomnia (Psychiatric disorders) | 6 | 8 | 10 | 8 | 3 | 4
Breast pain (Reproductive system and breast disorders) | 4 | 7 | 8 | 6 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 9 | 8 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 4 | 4 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 9 | 4 | 3 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 5 | 1 | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 8 | 7 | 10 | 4 | 9
Onychoclasis (Skin and subcutaneous tissue disorders) | 5 | 3 | 6 | 4 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 12 | 15 | 10 | 1 | 8
Hot flush (Vascular disorders) | 8 | 6 | 17 | 7 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT02400476/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02400476/SAP_001.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02400476/ICF_002.pdf